CLINICAL TRIAL: NCT06729983
Title: Prophylactic Conjoint Tendon Lengthening During Reverse Shoulder Arthroplasty: is There a Difference in Anterior Shoulder Pain At One Year After Surgery?
Brief Title: Prophylactic Conjoint Tendon Lengthening During Reverse Shoulder Arthroplasty Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nickolas Garbis (Other)
Collaborators: Loyola University School of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Nickolas Garbis, Chief of Shoulder/Elbow Division, Loyola University
Organization: Loyola University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 218607
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis Shoulder
Keywords: reverse shoulder athroplasty; conjoint tendon lengthening; pain outcome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Standard reverse shoulder arthroplasty
  Interventions: Procedure: Standard Reverse Shoulder Arthroplasty
- Treatment (Experimental): Prophylactic conjoint tendon lengthening in addition to reverse shoulder arthroplasty
  Interventions: Procedure: Prophylactic Conjoint Tendon Lengthening

INTERVENTIONS:
Procedure: Prophylactic Conjoint Tendon Lengthening — During a standard reverse shoulder arthroplasty procedure, the conjoint tendon will be incised and lengthened prophylactically
  Arms: Treatment
Procedure: Standard Reverse Shoulder Arthroplasty — A standard reverse shoulder arthroplasty procedure will be performed
  Arms: Control

SUMMARY:
Some patients may experience persistent pain in the front of their shoulder after reverse shoulder replacement. One of the possible reasons for this is that the surgery causes a change in the alignment of the shoulder joint, which may cause increased tension and compression on one of the biceps tendon called the conjoint tendon. The purpose of this study is to evaluate whether conjoint tendon lengthening, a surgical procedure that involves cutting and lengthening the conjoint tendon in order to reduce tension and compression, is able to prevent or reduce the risk of anterior shoulder pain at one year after surgery.

DETAILED DESCRIPTION:
Reverse shoulder arthroplasty (RSA) is a surgical procedure that is used to treat severe shoulder arthritis with rotator cuff damage. RSA involves reversing the ball and socket of the shoulder joint, such that the ball is attached to the shoulder blade and the socket is attached to the upper arm bone. This allows the deltoid muscle to take over the function of the rotator cuff and provide more stability and mobility to the shoulder. RSA has been shown to improve pain, function, and quality of life in patients with various shoulder conditions, such as rotator cuff tear arthropathy, glenohumeral osteoarthritis, complex proximal humeral fractures, pseudoparalysis, and revision shoulder arthroplasty.

However, some patients may experience persistent anterior shoulder pain after RSA, which can limit their function and quality of life. The exact cause and prevalence of this complication are not well understood, but several possible mechanisms have been proposed, such as impingement, instability, infection, nerve injury, fracture, scapular notching, and conjoint tendinitis.

Conjoint tendinitis is a condition where the tendon that connects the coracoid process to the upper arm bone, called the conjoint tendon, becomes inflamed and painful. The conjoint tendon is part of the biceps muscle and the coracobrachialis muscle, and it plays a role in shoulder flexion and internal rotation. Conjoint tendinitis may occur after RSA due to the increased tension and compression on the anterior shoulder caused by the shift in the center of rotation of the joint. Conjoint tendinitis may manifest as anterior shoulder pain, tenderness over the coracoid process, and decreased range of motion and strength.

Conjoint tendon lengthening (CTL) is a surgical procedure that involves cutting or lengthening the conjoint tendon, which may relieve the pain by reducing the tension and compression on the anterior shoulder. CTL can be performed as a primary procedure during RSA, or as a secondary procedure after RSA. The rationale for performing CTL as a primary procedure is to prevent the development of conjoint tendinitis and anterior shoulder pain after RSA. The rationale for performing CTL as a secondary procedure is to treat the patients who have failed conservative treatments, such as physical therapy, injections, or medications, and have persistent anterior shoulder pain after RSA.

The literature on CTL for anterior shoulder pain after RSA is scarce and mostly consists of case reports and case series. There is no randomized controlled trial or systematic review on this topic. The existing studies have reported favorable results of CTL, with improvement in pain, function, and patient-reported outcomes. However, the studies have also acknowledged the limitations of their methods, such as small sample size, lack of control group, short follow-up, and potential bias. Therefore, the evidence for the effectiveness of CTL for anterior shoulder pain after RSA is weak and inconclusive.

The gap or problem that this research aims to address is the lack of high-quality evidence on the effectiveness of prophylactic CTL during RSA for preventing or reducing anterior shoulder pain at one year after surgery. The investigators hypothesize that patients who undergo prophylactic CTL during RSA will have less anterior shoulder pain at one year after surgery than those who do not. The investigators will test this hypothesis by conducting a randomized controlled trial with two groups: CTL group and control group. The investigators will compare the pain intensity, range of motion, strength, activity level, and patient-reported outcomes of the two groups at 6 months and 12 months after RSA. The investigators will also identify the factors that predict the response to CTL, such as age, gender, body mass index, comorbidities, duration of pain, and severity of arthritis. This research will contribute to the knowledge in the field of shoulder surgery by providing high-quality evidence on the effectiveness of prophylactic CTL during RSA for anterior shoulder pain. This research will also have practical implications for the field of shoulder surgery by providing a viable option for patients who suffer from anterior shoulder pain after RSA, and enhancing their function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years old undergoing primary reverse total shoulder arthroplasty
* Operations that occur at Loyola University Medical Center (Maywood, IL), Loyola Ambulatory Surgery Center (Maywood, IL), or Gottlieb Memorial Hospital

Exclusion Criteria:

* Patients younger than 18 years old
* Patients who had prior coracoid transfer procedure
* Patients who are undergoing revision surgery from a prior arthroplasty
* Current pregnancy As per standard protocol with all surgeries, a urine pregnancy test is performed prior to surgery. If positive, the surgery will be cancelled and the patient will be excluded from the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
American Society of Shoulder and Elbow Surgeons (ASES) Score | From enrollment to the end of treatment at 12 months
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points. The higher the points the better the outcome.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | From enrollment to the end of treatment at 12 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10).
The Shoulder Pain and Disability Index (SPADI) | From enrollment to end of treatment at 12 months
  The Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with ADLs requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items. The patient is instructed to choose the number that best describes their level of pain and extent of difficulty using the involved shoulder. The pain scale is summed up to a total of 50 while the disability scale sums up to 80. The total SPADI score is expressed as a percentage. A score of 0 indicates best 100 indicates worst. A higher score shows more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Nickolas G Garbis, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola Outpatient Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This is a single cite study

REFERENCES:
- [Background] Werner BC, Chang B, Nguyen JT, Dines DM, Gulotta LV. What Change in American Shoulder and Elbow Surgeons Score Represents a Clinically Important Change After Shoulder Arthroplasty? Clin Orthop Relat Res. 2016 Dec;474(12):2672-2681. doi: 10.1007/s11999-016-4968-z. Epub 2016 Jul 8. PMID 27392769
- [Background] Vij N, Tummala S, Shahriary E, Tokish J, Martin S. Total Shoulder Arthroplasty Versus Reverse Shoulder Arthroplasty in Primary Glenohumeral Osteoarthritis With Intact Rotator Cuffs: A Meta-Analyses. Cureus. 2024 Apr 8;16(4):e57866. doi: 10.7759/cureus.57866. eCollection 2024 Apr. PMID 38725735
- [Background] Gomez GV, Huffman GR. Conjoint tendon lengthening for recalcitrant anterior shoulder pain after reverse shoulder arthroplasty: a technique article. JSES Rev Rep Tech. 2022 Jan 13;2(2):164-167. doi: 10.1016/j.xrrt.2021.12.005. eCollection 2022 May. PMID 37587959
- [Background] Tashjian RZ, Frandsen JJ, Christensen GV, Chalmers PN. Conjoint tendon release for persistent anterior shoulder pain following reverse total shoulder arthroplasty. JSES Int. 2020 Jul 31;4(4):975-978. doi: 10.1016/j.jseint.2020.07.005. eCollection 2020 Dec. PMID 33345243
- [Background] Boileau P, Melis B, Duperron D, Moineau G, Rumian AP, Han Y. Revision surgery of reverse shoulder arthroplasty. J Shoulder Elbow Surg. 2013 Oct;22(10):1359-70. doi: 10.1016/j.jse.2013.02.004. Epub 2013 May 22. PMID 23706884
- [Background] Black EM, Roberts SM, Siegel E, Yannopoulos P, Higgins LD, Warner JJ. Failure after reverse total shoulder arthroplasty: what is the success of component revision? J Shoulder Elbow Surg. 2015 Dec;24(12):1908-14. doi: 10.1016/j.jse.2015.05.029. Epub 2015 Jul 7. PMID 26163279
- [Background] Anakwenze OA, Kancherla VK, Carolan GF, Abboud J. Coracoid fracture after reverse total shoulder arthroplasty: a report of 2 cases. Am J Orthop (Belle Mead NJ). 2015 Nov;44(11):E469-72. PMID 26566565
- [Background] Schwartz DG, Kang SH, Lynch TS, Edwards S, Nuber G, Zhang LQ, Saltzman M. The anterior deltoid's importance in reverse shoulder arthroplasty: a cadaveric biomechanical study. J Shoulder Elbow Surg. 2013 Mar;22(3):357-64. doi: 10.1016/j.jse.2012.02.002. Epub 2012 May 19. PMID 22608931
- [Background] Schairer WW, Nwachukwu BU, Lyman S, Craig EV, Gulotta LV. National utilization of reverse total shoulder arthroplasty in the United States. J Shoulder Elbow Surg. 2015 Jan;24(1):91-7. doi: 10.1016/j.jse.2014.08.026. Epub 2014 Oct 29. PMID 25440519
- [Background] Kim SH, Wise BL, Zhang Y, Szabo RM. Increasing incidence of shoulder arthroplasty in the United States. J Bone Joint Surg Am. 2011 Dec 21;93(24):2249-54. doi: 10.2106/JBJS.J.01994. PMID 22258770
- [Background] Grammont PM, Baulot E. The classic: Delta shoulder prosthesis for rotator cuff rupture. 1993. Clin Orthop Relat Res. 2011 Sep;469(9):2424. doi: 10.1007/s11999-011-1960-5. No abstract available. PMID 21732025
- [Background] Drake GN, O'Connor DP, Edwards TB. Indications for reverse total shoulder arthroplasty in rotator cuff disease. Clin Orthop Relat Res. 2010 Jun;468(6):1526-33. doi: 10.1007/s11999-009-1188-9. PMID 20049573